CLINICAL TRIAL: NCT04894981
Title: Comparison of Power Wheelchair Driving Performance in a Physical Simulator With CAVE, Immersive Helmet and Non-immersive Screen in a Population of Drivers With Neurological Disorders: Pilot Study
Brief Title: Comparison of Power Wheelchair Driving Performance Under Immersive and Non-immersive Conditions With Drivers With Neurological Disorders
Acronym: SIMADAPT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Collaborators: INSA Rennes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-A00120-41
Record Dates: First submitted 2021-05-03; First posted 2021-05-20 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-05

CONDITIONS: Neurologic Disorder; Brain Injuries; Neurodegeneration
MeSH Terms: conditions — Nervous System Diseases; Brain Injuries; Nerve Degeneration | interventions — Early Detection of Cancer

STUDY DESIGN:
Intervention Model Description: This is a pilot, prospective, single-centre, controlled, randomised, crossover, open-label, study. (RIPH2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive condition (Experimental): Performance driving wheelchair in immersive condition (in Cave automatic environment or with HMD)
  Interventions: Device: Immersive condition (CAVE); Device: Immersive condition (HMD)
- Non Immersive condition (Experimental): Performance driving wheelchair in non immersive condition (with screen and physical simulator or screen only)
  Interventions: Device: Non Immersive condition (Screen alone); Device: Non Immersive condition (Screen with physical simulator)

INTERVENTIONS:
Device: Immersive condition (CAVE) — Driving course with obstacles in a CAVE system
  Arms: Immersive condition
Device: Immersive condition (HMD) — Driving course with obstacles with a virtual reality headset
  Arms: Immersive condition
Device: Non Immersive condition (Screen alone) — Driving course with obstacles on a screen with physical simulator
  Arms: Non Immersive condition
Device: Non Immersive condition (Screen with physical simulator) — Driving course with obstacles on a screen only
  Arms: Non Immersive condition

SUMMARY:
This study aims to assess the impact of the choice of visual feedback solution (immersive via CAVE and VR headset; non-immersive via screen only) on driving performance and quality of experience on a physical driving simulator and its acceptability to wheelchair drivers with neurological disorders.

DETAILED DESCRIPTION:
The device under investigation is an electric wheelchair driving simulation solution driving simulation solution for electric wheelchairs, based on a physical physical simulation device that integrates software allowing virtual virtual immersion. This device will be coupled with three visual simulation solutions: a virtual reality helmet, a CAVE (virtual reality room where video virtual reality room where video projectors display content on four sides) and a non-immersive projection (screen only, non-immersive virtual reality solution).

This device is intended to allow patients who may acquire a power wheelchair to train in a virtual environment, which is conducive to the safety of the training, its repetition, and to produce more varied training environments, richer and more adapted to specific and individualised needs. These solutions could facilitate access to real driving for patients who are currently experiencing learning difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 years of age,
* Patient with neurological disorders such as brain injury or neurodegeneration,
* Having been prescribed an electric wheelchair and circulating in electric wheelchair for more than 3 months
* Of which electric wheelchair is the main mode of travel
* Whose physical measurements (weight, height) are compatible with the use of the physical simulator chosen for the development of the robotic assistance module, i.e. according to the manufacturer's data 140 kg max and 51 cm max seat width.
* Having freely consented to participate in the study,
* In the case of curatorship, having read the patient information document and given his/her free and informed consent to participate in the study, in the presence of his/her curator,
* In the case of a guardianship, the legal representative having read the information document intended for the legal guardian of an adult under legal protection (under guardianship) and given his or her free and informed consent for the person for whom he or she is responsible to participate in the study (in agreement with the patient)

Exclusion Criteria:

* Comprehension problems that prevent the protocol from being carried out,
* Motor disorders of the upper limb requiring additional technical driving assistance,
* A patient who has expressed difficulties with internal and/or external driving safety on the basis of the WST,
* Patients who were included in the SIMADAPT1 study to avoid bias due to their experience in the simulator and virtual reality,
* Pregnant, parturient or breastfeeding women,
* Person deprived of liberty by a judicial or administrative decision, persons under psychiatric care or for purposes other than research,
* Minor,
* Person in emergency situation unable to give prior consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
number of the collisions with the environment on the standardised circuit | During the driving course, from the beginning to the end of the circuit.
  It will be compared in 4 conditions :
  * immersive 1: physical simulator and CAVE_condition A1
  * immersive 2: physical simulator and virtual reality helmet_condition A2
  * non-immersive 1: screen and physical simulator_condition B1
  * non-immersive 2: screen only without simulator_condition B2 Day 1 : A + B Day 8 : A + B

SECONDARY OUTCOMES:
the time taken to complete the course | During the driving course, from the beginning to the end of the circuit.
  It will be measured, in minutes and seconds, under the various conditions
evaluation of driving performance with Wheelchair Skill Test (WST-Q-T 5.1) | Immediately after intervention
  The Wheelchair Skill Test (WST-Q-T 5.1) will be completed by two evaluators after each condition.
  The score will be between 0 to 22, a high score will represent a good driving performance
visual information (VICON® system) | During the driving course, from the beginning to the end of the circuit.
  The number of head movement will be measured by VICON system.
the cognitive load of carrying out the circuit with National Aeronautics and Space Administration Task Load Index | Immediately after intervention
  The cognitive load of tests under each conditions will be measured by the NASA-Task Load Index. It is in the form of six scales where the participant must assign a score between zero and one hundred to each of them, score indicating a growing level of intensity. Three dimensions relate to the demands imposed on the subject (mental, physical and temporal demands) and three to the interaction of a subject with the task (effort, frustration and performance)
sensation of immersion and the feeling of presence in a virtual situation (Igroup Presence Questionnaire IPQ) | Immediately after intervention
  It will be evaluated and compared by Igroup Presence Questionnaire IPQ.
discomfort of driving in immersive reality, | Immediately after intervention
  The occurrence of kinetosis will be evaluated with Graybiel score by the two evaluators after each passage in each condition.
  The score is between 1 to 50. A high score shows the patient's discomfort.
satisfaction of the testers and the acceptability of the various conditions simulated | Immediately after intervention
  Patients will be asked to rate their satisfaction on a scale of 0 to 10, with 10 being very satisfied.
the acceptability of the various conditions simulated | Immediately after intervention
  Evaluation of acceptability with Unified Theory of Acceptance and Use of Technology (UTAUT) after each condition

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GALLIEN, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pole Saint-Hélier, Rennes, Brittany Region, France